CLINICAL TRIAL: NCT01210222
Title: A Phase II Trial of AMG 386, a Selective Angiopoietin 1/2 Neutralizing Peptibody, in Patients With Persistent/Recurrent Carcinoma of the Endometrium
Brief Title: Trebananib in Treating Patients With Persistent or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0229L; NCI-2011-02655 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000686066; GOG-0229L (Other: NRG Oncology); GOG-0229L (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2010-09-25; First posted 2010-09-28 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2017-08

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Adenosquamous Carcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Endometrioid Adenocarcinoma, Variant With Squamous Differentiation; Endometrial Serous Adenocarcinoma; Endometrioid Stromal Sarcoma; Recurrent Uterine Corpus Carcinoma
MeSH Terms: conditions — Sarcoma, Endometrial Stromal | interventions — trebananib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (trebananib) (Experimental): Patients receive trebananib IV over 30-60 minutes on days 1, 8, 15, and 21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Trebananib

INTERVENTIONS:
Biological: Trebananib — Given IV

SUMMARY:
This phase II trial studies the side effects and how well trebananib works in treating patients with persistent or recurrent endometrial cancer. Trebananib may stop the growth of endometrial cancer by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the proportion of patients with persistent or recurrent endometrial cancer, who survive progression-free for at least 6 months and the proportion of patients who have objective tumor response (complete or partial), treated with AMG 386 (trebananib).

II. To determine the nature and degree of toxicity of AMG 386 in this cohort of patients.

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival (PFS) and overall survival (OS) of patients with persistent or recurrent endometrial cancer treated with AMG 386.

OUTLINE:

Patients receive trebananib intravenously (IV) over 30-60 minutes on days 1, 8, 15, and 21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent endometrial carcinoma, which is refractory to curative therapy or established treatments; histologic confirmation of the original primary tumor is required; stained slides to document the primary tumor as well as recurrent/persistent disease (if documented by histology or cytology) are required
* Patients with the following histologic epithelial cell types are eligible:

  * Endometrioid adenocarcinoma
  * Serous adenocarcinoma
  * Undifferentiated carcinoma
  * Clear cell adenocarcinoma
  * Mixed epithelial carcinoma
  * Adenocarcinoma not otherwise specified (N.O.S.)
  * Mucinous adenocarcinoma
  * Squamous cell carcinoma
  * Transitional cell carcinoma
* All patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as 'non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence >= 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG phase III or Rare Tumor protocol for the same patient population
* Patients who have received one prior chemotherapy regimen must have a GOG performance status of 0, 1, or 2; patients who have received two prior chemotherapy regimens must have a GOG performance status of 0 or 1
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy
* Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI])
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
* Any other prior therapy directed at the malignant tumor, including chemotherapy and immunologic agents, must be discontinued at least three weeks prior to registration
* Any prior radiation therapy must be completed at least 4 weeks prior to registration
* Patients must have had one prior chemotherapeutic regimen for management of endometrial carcinoma; chemotherapy administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a chemotherapy regimen
* Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease
* Patients must have NOT received any non-cytotoxic (biologic or targeted) agents as part of their primary treatment or for management of recurrent or persistent disease

  * Non-cytotoxic (biologic or targeted) agents include (but are not limited to) monoclonal antibodies, cytokines, and small-molecule inhibitors of signal transduction
* Prior hormonal therapy is allowed; there is no limit on the number of prior hormonal therapies allowed
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Hemoglobin level >= 9.0 g/dL
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN) or a creatinine clearance >= 60 ml/m^2
* Bilirubin less than or equal to 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Neuropathy (sensory and motor) less than or equal to grade 1
* Prothrombin time (PT) such that international normalized ratio (INR) is =< 1.5 x ULN (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin) and a partial thromboplastin time (PTT) =< 1.5 x ULN
* Albumin >= 2.8 mg/dL
* Patients must have a urine protein of =< 1 on dipstick; if dipstick is 2+ or higher, 24-hour urine protein must be obtained and should be < 1 g for patient to be eligible
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients of child bearing potential must agree to use an accepted and effective non-hormonal method of contraception i.e., double barrier method (e.g. condom plus diaphragm) from the time of signing the informed consent through 6 months after last dose of study drug

Exclusion Criteria:

* Patients who are currently or have been previously treated with trebananib, or other molecules that inhibit the angiopoietins or Tie2 receptor
* Patient with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies, are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of endometrial cancer within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of endometrial cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients who are pregnant or nursing
* Patients with symptoms of partial or complete bowel obstruction; recent (within 6 months) history of fistula, intraabdominal abscess or bowel perforation; subjects requiring total parenteral nutrition or parenteral hydration
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including brain tumor, seizures not controlled with standard medical therapy or any brain metastases
* Patients with clinically significant cardiovascular disease; this includes:

  * Myocardial infarction or unstable angina within 12 months of the first date of study treatment
  * New York Heart Association (NYHA) Class II or greater congestive heart failure
  * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) or cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with anti-arrhythmic medication)
  * Grade 2 or greater peripheral vascular disease
  * Cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of study treatment
  * History of arterial ischemia or thrombus
* Patients with uncontrolled hypertension defined as systolic > 150 mm Hg or diastolic > 90 mm Hg; the use of anti-hypertensive medications to control hypertension is permitted
* Patients with significant bleeding within 6 months of enrollment or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients who have undergone major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to the first date of study treatment or who have major surgical procedure anticipated during the course of the study
* Patients who have undergone minor surgical procedures within 7 days of the first date of study treatment

  * Paracentesis and thoracentesis are permitted prior to and while on study at the discretion of the investigator and as clinically indicated
* Patients treated with immune modulators such as systemic cyclosporine or tacrolimus within 30 days prior to enrollment
* Patients with serious non-healing wound, ulcer (including gastrointestinal), or bone fracture
* Patients with known human immunodeficiency virus (HIV), hepatitis C or chronic or active hepatitis B
* Patients with any condition which, in the investigator's opinion, makes the patient unsuitable for study participation
* Patients not available for follow-up assessments
* Patients with known sensitivity to any of the products to be administered during dosing
* Patients with history of allergic reactions to bacterially produced proteins
* Patients with a history of venous or arterial thromboembolism within 12 months prior to enrollment/randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-06-06 (Actual); Primary Completion 2016-07-16 (Actual); Study Completion 2016-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Moore, Principal Investigator — NRG Oncology
Locations (33):
- United States (33):
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Memorial University Medical Center, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - University of Mississippi Medical Center, Jackson, Mississippi
  - CoxHealth South Hospital, Springfield, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: GOG 0229L accrued 35 patients from June 2011 to August 2012. 32 of these patients were eligible.
Period: Overall Study
Arm/Group | Treatment (Trebananib)
Started | 35
Completed | 32
Not Completed | 3
Not completed — Ineligible | 2
Not completed — Never treated | 1

BASELINE CHARACTERISTICS:
Population: Eligible and evaluable patients
Arm/Group | Treatment (Trebananib)
Number analyzed (Participants) | 32
Age, Customized [Count of Participants; unit: Participants]
  40 - 49 years | 1
  50 - 59 years | 6
  60 - 69 years | 11
  70 - 79 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival > 6 Months
Description: Whether or not the patient survived progression-free for at least 6 months.
Time Frame: At 6 months
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Trebananib)
Number analyzed (Participants) | 32
percentage of participants | 18.8 [8.5 to 33.7]

2. Primary Outcome: Objective Tumor Response (Complete or Partial Response)
Description: Complete and Partial Tumor Response by RECIST 1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 5 years
Population: Eligible and treated patients.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Trebananib)
Number analyzed (Participants) | 32
percentage of participants | 3.1 [0.2 to 14.0]

3. Primary Outcome: Adverse Events as Assessed by NCI CTCAE v 4.0
Time Frame: Up to 5 years
Population: Eligible and evaluable patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 4.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 4.0
- Grade 2 (CTCAE v 4.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 4.0
- Grade 3 (CTCAE v 4.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 4.0
- Grade 4 (CTCAE v 4.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 4.0
- Grade 5 (CTCAE v 4.0): Number of patients who experienced a grade 5 event using common terminology criteria version 4.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 4.0) | Grade 2 (CTCAE v 4.0) | Grade 3 (CTCAE v 4.0) | Grade 4 (CTCAE v 4.0) | Grade 5 (CTCAE v 4.0)
Number analyzed (Participants) | 32 | 32 | 32 | 32 | 32 | 32
Participants
  Fatigue | 10 | 11 | 9 | 2 | 0 | 0
  Anemia | 15 | 15 | 2 | 0 | 0 | 0
  Constipation | 16 | 10 | 6 | 0 | 0 | 0
  Hypertension | 20 | 1 | 7 | 4 | 0 | 0
  Nausea | 20 | 6 | 2 | 4 | 0 | 0
  Abdominal Pain | 20 | 1 | 3 | 8 | 0 | 0
  Edema Limbs | 21 | 4 | 5 | 2 | 0 | 0
  Anorexia | 22 | 6 | 3 | 1 | 0 | 0
  Peripheral Sensory Neuropathy | 22 | 10 | 0 | 0 | 0 | 0
  Cough | 24 | 7 | 1 | 0 | 0 | 0
  Diarrhea | 24 | 6 | 2 | 0 | 0 | 0
  Hyperglycemia | 24 | 6 | 2 | 0 | 0 | 0
  Hyponatremia | 24 | 5 | 0 | 2 | 1 | 0
  Hypoalbuminemia | 24 | 3 | 3 | 2 | 0 | 0
  Dyspnea | 25 | 4 | 1 | 2 | 0 | 0
  Vomiting | 25 | 2 | 3 | 2 | 0 | 0
  Ascites | 27 | 0 | 2 | 3 | 0 | 0
  Bloating | 28 | 1 | 3 | 0 | 0 | 0
  Lymphedema | 28 | 1 | 1 | 2 | 0 | 0
  Thromboembolic Event | 28 | 0 | 2 | 2 | 0 | 0
  Localized Edema | 29 | 3 | 0 | 0 | 0 | 0

4. Secondary Outcome: Overall Survival
Description: The observed length of life from entry into the study to death or the date of last contact.
Time Frame: From study entry to death or last contact, up to 5 years
Population: Eligible and treated patients
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Treatment (Trebananib)
Number analyzed (Participants) | 32
Months | 6.6 [4.01 to 14.75]

5. Secondary Outcome: Progression-free Survival
Description: The time from entry until disease progression, death, or date of last contact. Endpoints are progression or death. Patients who are not observed with an endpoint are censored. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Patients whose disease can be evaluated by physical exam, progression was assessed prior to each cycle. CT or MRI if used to follow leasion for measurable disease, up to 5 years
Population: Eligible and treated patients
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Treatment (Trebananib)
Number analyzed (Participants) | 32
Months | 2.0 [1.77 to 2.10]

ADVERSE EVENTS:
Time Frame: AEs were collected during treatment and up to 30 days after study treatment ended. Also reported are serious adverse events (SAEs) considered to be treatment related for up to 5 years after stopping study treatment.
Arm/Group | Treatment (Trebananib)
Serious Adverse Events (participants affected / at risk) | 14/32
Other Adverse Events (participants affected / at risk) | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trebananib) (N=32)
Colonic Obstruction (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 4
Abdominal Distension (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Edema Limbs (General disorders) | 1
Death Nos (General disorders) | 3
Kidney Infection (Infections and infestations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Seizure (Nervous system disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic Event (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Trebananib) (N=32)
Anemia (Blood and lymphatic system disorders) | 17
Palpitations (Cardiac disorders) | 2
Sinus Tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hearing Impaired (Ear and labyrinth disorders) | 1
Eye Disorders - Other (Eye disorders) | 1
Watering Eyes (Eye disorders) | 1
Flashing Lights (Eye disorders) | 1
Blurred Vision (Eye disorders) | 1
Eyelid Function Disorder (Eye disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 6
Dry Mouth (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 16
Diarrhea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 7
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 4
Abdominal Pain (Gastrointestinal disorders) | 9
Mucositis Oral (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Oral Cavity Fistula (Gastrointestinal disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 12
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2
Rectal Pain (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 1
Pain (General disorders) | 3
Localized Edema (General disorders) | 3
Irritability (General disorders) | 1
Flu Like Symptoms (General disorders) | 1
Edema Trunk (General disorders) | 1
Edema Limbs (General disorders) | 10
Edema Face (General disorders) | 1
Fatigue (General disorders) | 22
Fever (General disorders) | 1
Chills (General disorders) | 2
Urinary Tract Infection (Infections and infestations) | 2
Bronchial Infection (Infections and infestations) | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Wound Complication (Injury, poisoning and procedural complications) | 1
Investigations - Other (Investigations) | 1
Weight Loss (Investigations) | 2
Weight Gain (Investigations) | 3
Platelet Count Decreased (Investigations) | 3
Lymphocyte Count Decreased (Investigations) | 1
Inr Increased (Investigations) | 3
Hemoglobin Increased (Investigations) | 1
Ggt Increased (Investigations) | 2
Creatinine Increased (Investigations) | 3
White Blood Cell Decreased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 2
Alkaline Phosphatase Increased (Investigations) | 7
Alanine Aminotransferase Increased (Investigations) | 1
Activated Partial Thromboplastin Time Prolonged (Investigations) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hypercalcemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 10
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 10
Peripheral Motor Neuropathy (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Movements Involuntary (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Facial Muscle Weakness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Cognitive Disturbance (Nervous system disorders) | 1
Suicidal Ideation (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 4
Hallucinations (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 4
Anxiety (Psychiatric disorders) | 6
Agitation (Psychiatric disorders) | 1
Urinary Urgency (Renal and urinary disorders) | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 2
Urinary Incontinence (Renal and urinary disorders) | 1
Urinary Tract Pain (Renal and urinary disorders) | 3
Urinary Frequency (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 4
Hematuria (Renal and urinary disorders) | 3
Acute Kidney Injury (Renal and urinary disorders) | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1
Vaginal Dryness (Reproductive system and breast disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 2
Vaginal Discharge (Reproductive system and breast disorders) | 1
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Thromboembolic Event (Vascular disorders) | 4
Phlebitis (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 3
Hypertension (Vascular disorders) | 12
Hot Flashes (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less